CLINICAL TRIAL: NCT01791530
Title: International Multicenter Study of Ventilator Associated Tracheobronchitis.
Acronym: TAVeM
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Ignacio Martin-Loeches, MD PhD, Corporacion Parc Tauli
Other Study IDs: TAVeM
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Incidence of VAT
Keywords: VAT; VAP; Transition from VAT to VAP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MV>48h: 10-20 consecutive admissions with a predictive duration of intubation and mechanical ventilation > 48h.

SUMMARY:
Justification and background Ventilator-associated complications (VACs) are those complications that develop during a period of intubation of a patient . Pneumonia is the second most frequent infectious complication in the hospital, and ranks first in ICU, whose risk is increased more than 20 times by the presence of invasive mechanical ventilation and is called ventilator-associated pneumonia (VAP) . Whereas the information published regarding VAP in terms of diagnosis, treatment and impact on the outcome of critically ill patients is enormous.Ventilator-associated tracheobronchitis (VAT) incidence is lacking and complicated in part, since the definition remains controversial. In addition, the significance of tracheobronchial colonization as a risk factor for subsequent lower respiratory tract infection remains unclear . The upper and lower airways can become colonized . Several factors have been taken into account and do not differ from those involved in VAT and VAP development in patients under mechanical ventilation.

Definition VAT diagnosis is controversial and represents an actual problem in order to define the real incidence of VAT , There is currently no valid, reliable definition for VAT, and even the most widely-used VAT criteria and definitions are neither sensitive nor specific. The diagnosis of VAT is considered when a patient under invasive mechanical ventilation starts with fever, leukocytosis and new or increased purulent secretions by the endotracheal tube. A particular difficulty with much commonly used VAT definition (in order to distinguish from VAP) is the key point of the absence of pulmonary consolidation. Evidence suggests that chest radiograph findings do not accurately role out VAP. A taskforce on hospital-acquired pneumonia, and VAP has been recently published (European Respiratory Society (ERS), European Society of Clinical Microbiology and Infectious Diseases (ESCMID) and European Society of Intensive Care Medicine (ESICM)). Nosocomial tracheobronchitis definition includes occurrence of purulent tracheal secretion after ≥48 h of hospitalisation or mechanical ventilation plus ≥2 of the following: fever (≥38.5°C) or hypothermia (<36°C), leukocytosis (≥12 × 109/L), significant bacteriologic counts in respiratory secretions (≥103 cfu/mL for protected brush specimen (PBS) and ≥105 cfu/mL for endotracheal aspirates); absence of new pulmonary infiltrates compatible with pneumonia and absence of other causes of fever are mandatory. This definition needs to be further validated and can overdiagnose the incidence of VAT (and overuse of antibiotics) because the positive culture of respiratory secretions is not a mandatory item RATIONALE Given the possible high incidence of VAT, and its importance as a risk factor for VAP, and a potential target to treat in order to reduce VAP incidence, a large multicentre

DETAILED DESCRIPTION:
METHODS This prospective international multicentre observational study will be conducted in 8 countries ((Spain, France, Portugal, Brazil, Argentina, Ecuador, Bolivia and Colombia).) Inclusion criteria 10-20 consecutive admissions with a predictive duration of intubation and mechanical ventilation > 48h.

Exclusion criteria Predicted duration of intubation and mechanical ventilation ≤ 48h. Tracheostomy at ICU admission. Primary objective To determine the incidence of VAT in patients requiring intubation and mechanical ventilation >48h.

Secondary objectives To determine risk factors for VAT. To determine incidence and risk factors for transition from VAT to VAP. To determine microorganisms associated with VAT. To determine the impact of VAT on outcome.

ELIGIBILITY:
Inclusion Criteria:

* 10-20 consecutive admissions with a predictive duration of intubation and mechanical ventilation > 48h.

Exclusion Criteria:

* Predicted duration of intubation and mechanical ventilation ≤ 48h.
* Tracheostomy at ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10-20 consecutive admissions with a predictive duration of intubation and mechanical ventilation > 48h.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of VAT in patients requiring intubation and mechanical ventilation >48h. | 1 year
  To determine the incidence of VAT in patients requiring intubation and mechanical ventilation >48h.

SECONDARY OUTCOMES:
Secondary Objectives | 1 year
  To determine risk factors for VAT.
To determine incidence and risk factors for transition from VAT to VAP. | 1 year
To determine microorganisms associated with VAT. | 1 year
To determine the impact of VAT on outcome. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Martin-Loeches, MD PhD, Principal Investigator — CORPORACIÓ SANITÀRIA I UNIVERSITARIA PARC TAULÍ - HOSPITAL DE SABADELL
Locations (8):
- Argentina, Argentina, Argentina
- Bolivia, Bolivia, Bolivia
- Brazil, Brazil, Brazil
- Colombia, Colombia, Colombia
- Ecuador, Ecuador, Ecuador
- France, France, France
- Portugal, Portugal, Portugal
- Corporació Sanitària I Universitaria Parc Taulí - Hospital de Sabadell, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Martin-Loeches I, Torres A, Povoa P, Zampieri FG, Salluh J, Nseir S, Ferrer M, Rodriguez A; TAVeM study Group. The association of cardiovascular failure with treatment for ventilator-associated lower respiratory tract infection. Intensive Care Med. 2019 Dec;45(12):1753-1762. doi: 10.1007/s00134-019-05797-6. Epub 2019 Oct 16. PMID 31620836
- [Derived] Martin-Loeches I, Povoa P, Rodriguez A, Curcio D, Suarez D, Mira JP, Cordero ML, Lepecq R, Girault C, Candeias C, Seguin P, Paulino C, Messika J, Castro AG, Valles J, Coelho L, Rabello L, Lisboa T, Collins D, Torres A, Salluh J, Nseir S; TAVeM study. Incidence and prognosis of ventilator-associated tracheobronchitis (TAVeM): a multicentre, prospective, observational study. Lancet Respir Med. 2015 Nov;3(11):859-68. doi: 10.1016/S2213-2600(15)00326-4. Epub 2015 Oct 22. PMID 26472037